CLINICAL TRIAL: NCT00028626
Title: Clinical Efficacy And Biologic Effects Of Preoperative Portal Vein Embolization In Patients With Colorectal Liver Metastases
Brief Title: Portal Vein Embolization in Treating Patients With Liver Metastases From Primary Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-113; CDR0000069112 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-2039
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Embolization, Therapeutic

INTERVENTIONS:
Drug: embolization therapy

SUMMARY:
RATIONALE: Embolization blocks blood flow to part of an organ and/or tumor. Blocking the portal vein on one side of the liver may cause the opposite side of the liver to increase in size and decrease the risk of liver failure following surgery.

PURPOSE: Phase II trial to study the effectiveness of portal vein embolization in treating patients who have liver metastases from primary colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether portal vein embolization results in significant hypertrophy of the remaining liver and potentially decreases the risk of liver failure after hepatic resection in patients with liver metastases from primary colorectal cancer.
* Determine the biologic effects of this therapy on liver metastases and normal liver parenchyma in these patients.

OUTLINE: Patients undergo portal vein embolization with 200-300 micron polyvinyl chloride particles suspended in Iohexol 300. Approximately 3-6 weeks after embolization, patients undergo an exploratory laparotomy followed by hepatic surgical resection.

Patients are followed for at least 6 months.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary colorectal adenocarcinoma with metastases to the liver being considered for hepatic resection
* Requirement for removal of at least 60% of functional liver parenchyma based on CT scan
* No extrahepatic disease by laparoscopy

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.8 mg/dL
* AST and ALT no greater than 80 IU/L

Renal:

* Creatinine no greater than 1.8 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 1 month since prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* At least 2 months since prior investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald DeMatteo, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States